CLINICAL TRIAL: NCT06209671
Title: A Clinical Study to Evaluate the Safety and Efficacy of INS19 CAR-T Cells for the Treatment of Relapsed or Refractory Acute B Lymphoblastic Leukemia
Brief Title: INS19 CAR-T Cells for the Treatment of Relapsed or Refractory Acute B Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1901
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Leukemia, B-cell
Keywords: INS19 CAR-T; Acute B-lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INS19 CAR-T Cells (Experimental): After preconditioning with chemotherapy, INS19 CAR-T Cells will be evaluated
  Interventions: Biological: INS19 CAR-T Cells

INTERVENTIONS:
Biological: INS19 CAR-T Cells — INS19 CAR-T Cells, 1-2×10^7 cells, treatment follows a lymphodepletion. Drug: Fludarabine Recommendation: 25-30 mg/m^2/day (D-5~D-3), determined by tumor burden at baseline. Drug: Cyclophosphamide Recommendation: 250-300 mg/m^2/day (D-5~D-3), determined by tumor burden at baseline.

SUMMARY:
This study, a single-center, open, single-dose clinical study, was designed to evaluate the safety, tolerability, and pharmacokinetic profile of INS19 CAR-T cells for the treatment of patients with relapsed or refractory acute B lymphoblastic leukemia

DETAILED DESCRIPTION:
The study is planned to enroll 9-12 patients with relapsed or refractory acute B-lymphoblastic leukemia in a modified "3+3" design with two dose groups of 1×10^7 cells and 2×10^7 cells (dose halved for subjects weighing <40 kg). Each dose group is planned to enroll 3-6 subjects to assess safety, and ultimately the SRC will decide whether to continue to add escalating dose groups or to conduct an extension study in a specific dose group based on available safety and efficacy information, with 3-6 subjects to be enrolled in the extension phase.

This study will be divided into a screening period, a cell collection period, a chemotherapy pretreatment period, a return infusion and a follow-up period, and within 28 days of return infusion the investigator will assess whether a DLT (Dose limited toxicity) event has occurred to confirm the safety of this dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory acute B-lymphoblastic leukemia who meet one of the following criteria and are diagnosed as CD19 positive by flow cytometry or histology, with the following provisions for the patient's prior treatment:

1. 2 or more bone marrow relapses;
2. Chemoresistance: relapse after chemotherapy and failure to achieve complete remission (MRD >1%) with at least 1 additional course of chemotherapy;
3. Relapse after autologous or allogeneic hematopoietic stem cell transplantation: time from transplantation to reinfusion is at least greater than 6 months;
4. Primary refractory: complete remission not achieved after two courses of standard chemotherapy (MRD >1%); 2. Philadelphia chromosome-positive (Ph+) patients are required to meet the following criteria: they should have received at least one relapse or refractory treatment with a tyrosine kinase inhibitor (TKI) agent ± chemotherapy or be intolerant of relapse or refractory to treatment with a TKI analog ± chemotherapy; Ph+ acute lymphoblastic leukemia (ALL) known to be accompanied by a T315I mutation, in the absence of an effective treatment with a TKI analog, is not require patients to be treated with TKI analogs ± chemotherapy; 3. Patients must have evaluable evidence of disease (bone marrow morphology suggestive of ≥5% primitive naive cells or bone marrow MRD >1%); 4. Age 3-70, including boundary values; 5. Expected survival of 3 months or more; 6. Eastern Cooperative Oncology Group (ECOG) score of 0-1 for patients aged 16 years and older (refer to Attachment 1); Lansky score of >50 for patients under 16 years of age (refer to Attachment 2); 7. Women of childbearing potential who have a negative blood pregnancy test prior to the start of the trial and who agree to use effective contraception for the duration of the trial until the last follow-up visit; male subjects whose partners are of childbearing potential agree to use effective contraception for the duration of the trial until the last follow-up visit; 8. Blood cell analysis meet the requirement 9. Adequate organ function 10. Toxicity due to prior therapy has stabilized or recovered to ≤ grade 1 or is not considered clinically significant by the investigator; 11. Volunteer to participate in this trial and sign on the informed consent

Exclusion Criteria:

1. Isolated extramedullary disease relapse;
2. Leukemia patients with symptoms of significant central nervous system invasion and requiring targeted therapy;
3. Prior treatment with a gene product;
4. Plasmapheresis with symptoms of compression (e.g., pleural effusion, abdominal effusion);
5. Patients with cardiac involvement and gastrointestinal involvement;
6. Autoimmune disease requiring systemic immunosuppressive therapy (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) within 2 years prior to the start of screening;
7. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, active arrhythmia, or other clinically significant cardiac disease within 6 months prior to the start of screening; patients with NYHA scores greater than Class I (or is it Class II);
8. Patients with a history of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to the start of screening; or requiring long-term antiplatelet therapy; or undergoing anticoagulation therapy;
9. Allergy to the study drug and related ingredients (e.g., albumin);
10. Those with Graft-versus-host disease (GVHD) requiring immunosuppression; or GVHD ≥ grade 2 or on anti-GVHD therapy; use of any medication for the treatment of GVHD within 4 weeks prior to enrollment; or autoimmune disease;
11. Provisions for prior medication:

    1. Systemic therapy (including chemotherapy, TKI inhibitors, and belintuzumab) 1 week or 5 half-lives prior to the cell collection period; clofarabine or cladribine within 3 months prior to enrollment, or pembrolizumab within 3 weeks prior to enrollment;
    2. Those who have combined systemic steroid medications within 5 days prior to the cell collection period (except those who have recently or are currently using topical or inhaled steroids);
    3. Those who have used drugs to stimulate bone marrow hematopoietic cell production within 5 days prior to the cell collection period;
    4. Patients who have participated in another clinical study within 1 month prior to screening; or who are scheduled to participate in a clinical trial of another drug during this study; however, enrollment will be allowed if the treatment is ineffective or the disease has progressed during the trial and at least 5 half-lives have elapsed prior to cell collection;
    5. INS19 CAR-T cells have received allogeneic cell therapy, such as donor lymphocyte transfusion, within 6 weeks prior to transfusion;
    6. Prior CAR-T cell therapy;
    7. Prior treatment with anti-CD19 target (unless CD19 target test remains positive);
    8. If immunotherapy such as anti-PD1, PD-L1, etc. has been used prior to INS19 CAR-T cell infusion, at least 4 weeks must have elapsed after the last dose and prior to INS19 CAR-T cell infusion;
    9. Live vaccination within 6 weeks prior to the start of screening. ii;
12. Prior or clinically significant CNS disorders at screening, such as epilepsy, epileptic seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disorders, organic brain syndromes, or psychiatric disorders;
13. Patients has HBV, HCV, HIV ,EBV, CMV or syphilis infection at the time of screening;
14. Pregnant or lactating, or planning pregnancy within 180 days after the end of CAR-T cells infusion, or male patients whose partners plan pregnancy 180 days after their CAR-T cell infusion;
15. History of malignancy other than non-melanotic skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) (unless in a disease-free state for at least 5 years);
16. Infections (fungal, bacterial, viral, or other) that require intravenous antimicrobial control or are uncontrollable, for simple urinary tract infections, and for bacterial pharyngitis, if the investigator assesses that they can be controlled by curative treatment, are eligible for enrollment.
17. Comorbid hereditary bone marrow failure-related syndromes such as Fanconi anemia, Kostmann syndrome, Schwachman syndrome, or other bone marrow failure syndromes, except Down syndrome;
18. The presence of any factors affecting compliance with the protocol, or the unwillingness or inability of the subject to comply with the procedures required in the study protocol, as judged by the investigator.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 28 days after CAR-T cell infusion
  Incidence of adverse events associated with CAR-T treatment, abnormal clinically significant laboratory findings, including dose-limiting toxicity (DLT) and maximum-tolerated Dose (MTD).
Persistence of CAR-T cells | Up to 24 weeks after CAR-T cell infusion
  cell counts and cell percentage in peripheral blood and bone marrow

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 28 days, 3 months and 6 months after CAR-T cell infusion
  Objective response rate (ORR)
Relapse free survival (RFS) | At 28 days, 3 months and 6 months after CAR-T cell infusion
  Relapse free survival (RFS)
Relapse free survival (RFS) | Up to 24 months after CAR-T cell infusion
  Relapse free survival (RFS)
Duration of response (DOR) | Up to 24 months after CAR-T cell infusion
  Duration of response (DOR)
Overall survival (OS) | Up to 24 months after CAR-T cell infusion
  Overall survival (OS)
Minimal residual disease (MRD) negative rate | Up to 24 months after CAR-T cell infusion
  Minimal residual disease (MRD) negative rate
Minimal residual disease (MRD) negative duration | Up to 24 months after CAR-T cell infusion
  Minimal residual disease (MRD) negative duration
Anti-therapeutic INS19 CAR-T cells antibody | Up to 24 months after CAR-T cell infusion
  Anti-therapeutic INS19 CAR-T cells antibody

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Zhao, PhD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No